CLINICAL TRIAL: NCT01112462
Title: A Single-dose, Randomized, Crossover Bioequivalence Study to Compare Two Formulations of Paracetamol/Phenylephrine
Brief Title: To Test Bioequivalence Between Two Formulations of Paracetamol/Phenylephrine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SC02009; 2009-018093-55 (EudraCT Number)
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Respiratory Tract Infections
Keywords: Nasal congestion, Headache
MeSH Terms: conditions — Respiratory Tract Infections; Nasal Obstruction; Headache | interventions — Acetaminophen; Phenylephrine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablet (Experimental): Paracetamol 500 mg/Phenylephrine 5 mg tablet
  Interventions: Drug: Paracetamol 500 mg/Phenylephrine 5 mg tablets
- Sachet (Active Comparator): Paracetamol 1000 mg/Phenylephrine 10 mg sachet
  Interventions: Drug: Paracetamol 1000 mg/Phenylephrine 10 mg sachet

INTERVENTIONS:
Drug: Paracetamol 500 mg/Phenylephrine 5 mg tablets — 2 tablets to be administered orally with 240 ml of water with a 24 hour follow-up period
  Other Names: Sudafed PE Sinus Pain Relief™
  Arms: Tablet
Drug: Paracetamol 1000 mg/Phenylephrine 10 mg sachet — 1 sachet dissolved in 240 ml water and administered orally with a 24 hour follow-up period
  Other Names: Flu Plus Hot Lemon™ sachet
  Arms: Sachet

SUMMARY:
This study is designed to assess bioequivalence between two paracetamol/ phenylephrine combination products.

DETAILED DESCRIPTION:
The study will be a single dose, randomized, two-way crossover study in 40 healthy subjects, with equal numbers of males and females. Drop-outs will not be replaced. The two doses of medication given in the study (a single dose in each of the two study periods) will be separated by a washout period of at least 7 days. In each study period, sixteen blood samples for pharmacokinetic analysis will be taken over 24 hours. Blood samples will be centrifuged and concentrations of paracetamol and phenylephrine in plasma will be measured using a validated chromatographic assay. Pharmacokinetic parameters will be calculated from plasma concentration data. The rate and extent of absorption of the formulations will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female
* Caucasians
* Aged between 18 and 50 years
* BMI ≤ 30 kg/m2
* Clinically normal medical history
* Physical normal examination
* Normal laboratory test results

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy
* Hypersensitivity to or intolerant of the study medications
* Donation or loss of blood within 90 days preceding the first dose of study medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measurements | during 24 hours following drug administration
  Pharmacokinetic measurements including:
  * Cmax (Maximum concentration)
  * AUC0-t (Area under the plasma concentration versus time curve from 0h to the lastmeasurable concentration)
  * AUC0-inf (Area under the plasma concentration versus time curve from 0h to infinity)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Shandon Clinical Trials Ltd., Cork, Ireland